CLINICAL TRIAL: NCT07119892
Title: Lifestyle Intervention and Its Effects on Inflammatory Cytokines and Oxidative Stress Markers in Diabetic Chronic Kidney Disease Patients: A Randomized Controlled Trial
Acronym: Lifestyle Inte
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Amany Gomaa Atiaa, lecturer, Sinai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU.REC.2025(46H)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus; Inflammation, Chronic Low-Grade; Chronic Kidney Disease; Stage 3 Chronic Kidney Disease; Stage 4 Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Renal Insufficiency, Chronic | interventions — Exercise; Diet

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: single Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Modification Group (Intervention) (Experimental): Participants engaged in a 12-week supervised aerobic exercise program (5x/week) at 70% of max HR, plus a calorie-restricted Mediterranean-style diet (1,200 kcal/day). Weekly dietitian counseling included Ramadan adjustments.
  Interventions: Behavioral: Lifestyle Modification (Exercise + Diet)
- Standard Care Group (No Intervention): Participants received routine nephrology care without structured lifestyle changes.

INTERVENTIONS:
Behavioral: Lifestyle Modification (Exercise + Diet) — Participants received a 12-week supervised aerobic exercise program (5 sessions per week at 70% of age-predicted maximum heart rate) and dietary counseling with a calorie-restricted Mediterranean-style diet of 1,200 kcal/day. The intervention was culturally adapted, including modifications for Ramadan.
  Arms: Lifestyle Modification Group (Intervention)

SUMMARY:
This randomized controlled trial investigated the effects of a 12-week structured lifestyle intervention-including supervised aerobic exercise and a calorie-restricted diet-on inflammatory cytokines and oxidative stress biomarkers in overweight adults with type 2 diabetes mellitus (T2DM) and moderate chronic kidney disease (CKD stages 3-4). A total of 60 sedentary participants aged 36-58 years were randomly assigned to either the intervention group or the control group. The primary outcomes included changes in TNF-α, IL-6, and sCRP levels. Secondary outcomes assessed oxidative stress markers (MDA, CD) and antioxidant enzymes (GSH, SOD, GPx).

DETAILED DESCRIPTION:
Diabetic CKD is characterized by chronic low-grade inflammation and heightened oxidative stress, both of which contribute significantly to cardiovascular morbidity and kidney function decline. This study evaluated whether a 12-week structured lifestyle intervention could improve systemic inflammatory and oxidative profiles in overweight adults with T2DM and CKD stages 3-4. Participants in the intervention group underwent supervised aerobic exercise (5 sessions/week) and received individualized dietary counseling with a 1,200 kcal/day Mediterranean-style diet. The control group received standard nephrology care without lifestyle modification. Outcomes were measured pre- and post-intervention and included pro-inflammatory markers (TNF-α, IL-6, sCRP), lipid peroxidation markers (MDA, CD), and antioxidant defenses (GSH, SOD, GPx). The intervention group demonstrated statistically significant improvements in all biomarker categories compared to controls. The study supports the integration of structured lifestyle interventions into standard care for diabetic CKD patients to improve redox balance and reduce inflammatory burden.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following:

* Diagnosed with Type 2 Diabetes Mellitus (T2DM)
* Diagnosed with moderate chronic kidney disease (CKD Stage 3 or 4), with eGFR 25-60 mL/min/1.73 m²
* Age between 36 and 58 years
* BMI between 30-35 kg/m² (classified as obese)
* Sedentary lifestyle, defined as <30 minutes of physical activity per week over the past 6 months
* Stable medication regimen for at least 3 months
* Willing and able to provide informed consent

Exclusion Criteria:

* Participants will be excluded if they:
* Use anti-inflammatory medications regularly
* Have congestive heart failure (CHF) or coronary artery disease (CAD)
* Have moderate to severe valvular heart disease
* Have active liver disease (ALT > 3× upper normal limit)
* Have orthopedic limitations preventing exercise participation
* Are currently pregnant or lactating
* Have received a kidney transplant
* Have respiratory failure or chronic pulmonary disease
* Are smokers (current) Have participated in a lifestyle intervention trial within the last 6 months

Ages: 36 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 36 Years to 58 Years (Adult)
Enrollment: 60 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
TNF-α (pg/mL) | Baseline and Week 12
  Change in tumor necrosis factor-alpha
sCRP (mg/L) | Baseline and Week 12
  Change in serum C-reactive protein levels
IL-6 (pg/mL) | Baseline and Week 12
  Change in interleukin-6 levels

SECONDARY OUTCOMES:
MDA (mmol/L) | Baseline and Week 12
  Malondialdehyde levels (oxidative stress marker)
CD (mmol/L) | Baseline and Week 12
  Conjugated dienes levels
GSH (mmol/gHb) | Baseline and Week 12
  Reduced glutathione level
GPx (units/gHb) | Baseline and Week 12
  Glutathione peroxidase enzyme activity
SOD (units/mL) | Baseline and Week 12
  Superoxide dismutase activity
BMI (kg/m²) | Baseline and Week 12
  Body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Manshyet El-Bakry Hospital, Cairo, Egypt